CLINICAL TRIAL: NCT06799689
Title: EFFECT OF ESMADEM EDUCATION MODEL ON RELIGIOUS COPING, TOLERANCE AND DEPRESSION OF RISKY PREGNANTS
Brief Title: The Effect of Esmadem Education Model on Spiritual Coping, Tolerance and Depression of High-Risk Pregnant Women
Acronym: smadem Educati
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Mine Gokduman Keles, Principal Investigator, PhD midwife, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 08.01.2025/01/21decision no
Record Dates: First submitted 2025-01-15; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Pregnant Women
Keywords: pregnant women; spiritual; prenatal attachment; doğum korkusuna

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- ESMADEM EDUCATİON (Active Comparator)
  Interventions: Behavioral: esmadem education

INTERVENTIONS:
Behavioral: esmadem education — By providing information about Esma-i Husna, the journey of knowing oneself and character building with Esma-i Husna will be emphasized. It will be carried out with the aim of building on 99 names, namely Allah, Rahman and Rahim, and reducing depressive feelings by benefiting from the guidance of these names.In the second session, it will be explained through the names Esma-i Husna, Celal and Cemal in order to manage depressive feelings and contribute to positive coping. The togetherness of pain as well as happiness, ease along with difficulty, joy along with sadness in a balanced life will be discussed with the name "Zü'l Celâl ve'l İkram" and the study of "Journey to perfection through the names Celal and Cemal". The meaning of existence and life in spirit will be discussed through the name Rab, the life cycle will be explained by establishing a relationship with the names Hafıd-Râfi, Kâbıd-Bâsıt, Muız-Müzil. In addition, it will be carried out within the framework of the name Hakim,
  Arms: ESMADEM EDUCATİON

SUMMARY:
Pregnancy is a normal and natural process in a woman's life. During this process, anatomical, physiological, biochemical and emotional changes are observed. The changes are a period in which social, biophysical and psychological changes are experienced, which also means a journey into the unknown for the woman and her family. Although the scope of prenatal care is high today, the main focus is on the physical aspects of care and medical precautions. Midwives who provide holistic care should also address spiritual care. Therefore, the ESMADEM training model will be conducted to examine the effect of the spiritual coping, prenatal attachment and fear of birth of pregnant women.

DETAILED DESCRIPTION:
Pregnancy is a normal and natural process in a woman's life. During this process, anatomical, physiological, biochemical and emotional changes are observed. The changes are a period in which social, biophysical and psychological changes occur, which also mean a journey into the unknown for the woman and her family . It has been reported that supporting pregnant women by midwives during this period and encouraging birth as a positive experience reduces fear of birth and increases prenatal attachment . In facilitating adaptation to the changes experienced and increasing the level of health; Complementary practices and education such as exercise, biofeedback, meditation, and prayer are used . One of these practices is spiritual care. Spirituality involves recognizing one's goals in life and the meaning of life. These conceptualizations are not always associated with religious beliefs. The purpose of spiritual care is to help people seek meaning and purpose in life. Spiritual teachings can have behavioral, cognitive, emotional and ethical aspects and can manifest themselves with trust, patience and prayer . One of these prayers is Esmâ-i Hüsnâ. Esmâ-i Hüsnâ is an expression that expresses all the names that are stated to belong to. Esmadem: It is a spiritual support model that provides significant contributions to spiritual development and life skills, where life skills are acquired and psychological and guidance practices are included, and aims at cognitive, emotional and behavioral gains. In this model, the name Şekur is taken as the center for stress. Along with this center name, the names Hallak, Bâki, Melik, Kahhâr and Muntekim are given for depression; Müheymin and Rakib for anxiety; and Halim, Latif, Rezzak, Rahman, Rahim for stress. Although the scope of prenatal care is high today, it is seen that the main focus is on the physical aspects of care and medical precautions. Midwives who provide holistic care should also take spiritual care into consideration. Therefore, the ESMADEM training model will be conducted to examine the effect of the spiritual coping, prenatal attachment and fear of birth of pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak, understand and write Turkish,
* Ages 18-35,
* Having a spontaneous pregnancy,

  * Volunteering to participate in the study,
  * According to the last menstrual period (LMS) or ultrasonography (USG) records, in the 24th week of pregnancy,
  * No risk factors,
  * Having a phone number to contact for educational meetings,
  * Participating in a pregnancy school

Exclusion Criteria:

* Pregnant women who had fear of childbirth

  * Chronic and/or psychiatric health problems
  * Failed to attend at least three sessions of the training program Who were at risk during any stage of the study Who could not be interviewed within the first 24 hours after birth were excluded from the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 96 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Religious Coping Scale | baseline and 3 months.
  Positive and negative religious coping scores are calculated separately in the scale. A total religious coping score is not obtained. The raw score that can be obtained from the positive religious coping subscale varies between 7 and 28, and the raw score that can be obtained from the negative religious coping subscale varies between 3 and 12.

IPD SHARING:
Plan to Share IPD: Yes